CLINICAL TRIAL: NCT01551368
Title: Using Nimodipine, a Calcium Channel Blocker, to Prevent the LH Surge and Ovulation in Women Undergoing Assisted Reproduction
Brief Title: Use of a Calcium Channel Blocker to Prevent Premature Luteinizing Hormone Surges in Infertility Patients
Acronym: nimodipine
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: small number of patients got recruited
Sponsor: Mount Sinai Hospital, Canada (Other)
Responsible Party: Principal Investigator, Robert Casper, Professor, Obstetrics and Gynecology, Mount Sinai Hospital, Canada
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 09-0175-A
Record Dates: First submitted 2011-12-15; First posted 2012-03-12 (Estimated); Last update posted 2019-03-08 (Actual); Status verified 2019-03

CONDITIONS: Infertility
Keywords: male factor; intrauterine insemination; LH surge; controlled ovarian stimulation; clomiphene citrate; letrozole; human menopausal gonadotropins
MeSH Terms: conditions — Infertility | interventions — Nimodipine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nimodipine (Experimental): Nimodipine 30 mg tablets will be self-administered by the subjects every 6 hours starting on the day that the ultrasound criterion for hCG triggering is met. The tablets will be taken for two days or until an LH surge is detected, whichever comes first. If no LH surge by 2 days, the hCG trigger (250 micrograms recombinant hCG) will be given followed by intrauterine insemination (IUI)in 40 hours. If the LH surge is detected, hCG will be given immediately and two IUIs will be performed 24 hours apart.
  Interventions: Drug: Nimodipine
- Placebo (Placebo Comparator): Same as for nimodipine but an identical placebo will be self-administered.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Nimodipine — Nimodipine 30 mg tablets will be self-administered by the subjects every 6 hours starting on the day that the ultrasound criterion for hCG triggering is met. The tablets will be taken for two days or until an LH surge is detected, whichever comes first. If no LH surge by 2 days, the hCG trigger (250 micrograms recombinant hCG) will be given followed by intrauterine insemination (IUI)in 40 hours. If the LH surge is detected, hcg will be given immediately and two IUIs will be performed 24 hours apart.
  Other Names: Nimotop
  Arms: Nimodipine
Drug: Placebo — Identical inactive tablets.
  Other Names: placebo tablets
  Arms: Placebo

SUMMARY:
Nimodipine (Nimotop® Bayer Pharmaceuticals Corporation), unlike other calcium channel blockers is fat soluble and therefore is able to cross the blood-brain barrier1. Gonadotropin releasing hormone (GnRH) neurons are clustered in the hypothalamus and are dependent on calcium flux to release GnRH responsible for the release of follicle-stimulating hormone (FSH) and luteinizing hormone (LH) from the anterior pituitary. In a natural menstrual cycle a spontaneous LH surge occurs mid-cycle which triggers ovulation. The investigators hypothesized that nimodipine, by blocking calcium channels, may effectively suppress the release of GnRH and consequently the natural LH surge.

In this prospective double-blinded randomized study the investigators will evaluate the efficacy of nimodipine to inhibit the natural LH surge in women undergoing controlled ovarian stimulation (COS) and intrauterine insemination (IUI). Nimodipine, if successful, may represent an inexpensive oral medication as an alternative to the currently used GnRH agonists or GnRH antagonists in assisted reproductive technologies like IVF.

DETAILED DESCRIPTION:
In reproductive aged women regular ovulatory cycles generate 1-2 mature ovarian follicles every month. Approximately mid-cycle a natural LH surge is observed and predictably induces ovulation within 24-36 hours. LH is a hormone produced by the anterior pituitary gland and is released in response to GnRH. Concurrently GnRH is synthesized and released in a pulsatile manner from GnRH neurons within the hypothalamus.

One of the essential steps of successful IVF is to ensure the properly timed aspiration of mature follicles from the ovaries prior to ovulation. If ovulation were to precede aspiration then the oocytes would have already been released and become unobtainable. Therefore inhibiting spontaneous ovulation is a crucial component of successful oocyte retrieval. In the clinical setting of IUI no oocyte retrieval is required, but appropriate timing of insemination with respect to ovulation is critical.

A premature LH surge and subsequent premature luteinization may occur in up to a third of ovarian stimulation cycles using gonadotropins (applicable to both IUI and IVF cycles), making it a major cause of treatment cancellation and having a negative impact on pregnancy outcomes 2-5. The most commonly used medications to prevent a premature LH surge are GnRH agonists and more recently GnRH antagonists. They are both commonly administered subcutaneously on a daily basis and act on the anterior pituitary gland (through different mechanisms) to inhibit the release of LH. Besides the additional patient cost and burden, these medications are associated with prolonged treatment protocols and decreased ovarian response to stimulation.

Nimodipine is a unique calcium channel blocker with lipophilic properties and a greater affinity for cerebral vasculature, and therefore has the ability to cross the blood-brain barrier. In a study on mice with induced intracerebral hemorrhage, nimodipine treatment improved cerebral bloodflow and displayed anti-ischemic effects. Nimodipine has obtained FDA approval to reduce the severity of neurological deficits in patients who have had a recent subarachnoid hemorrhage.

On a cellular level nimodipine has been shown to inhibit the pulsatile activity of GnRH gene expression, an intrinsic property of GnRH neurons that is necessary for proper initiation of the LH surge. Specifically, nimodipine blocks L-type voltage gated calcium channels which prevent the influx of extracellular calcium and subsequently the stimulation of GnRH release. The intrinsic pulsatile secretion of GnRH has been directly associated with the rhythmic changes in intracellular calcium concentration in GnRH neurons.

Study Objectives and Endpoints

Primary Objective

1. To determine if nimodipine can effectively inhibit the natural LH surge in women undergoing controlled ovarian stimulation and intrauterine insemination.

   Secondary Objectives
2. To determine the medication side effect profile of nimodipine, specifically symptoms of hypotension, tachycardia, nausea or headache.
3. To determine the treatment compliance rate (nimodipine or placebo).
4. To determine the clinical pregnancy rate for each intervention arm (nimodipine or placebo) during the COS and IUI treatment cycle.

Primary Endpoint

1. The presence or absence of an LH surge on intervention Day 1 and Day 2. LH surge will be determined by serum LH levels at least two times the baseline serum LH.

   Baseline serum LH = (Cycle Day 3 serum [LH] + Cycle Day 7 serum [LH]) /2.

   Secondary Endpoint
2. Medication side effect profile:

   * Symptomatic hypotension [Note: vital signs will not be routinely recorded]
   * Symptomatic tachycardia [Note: vital signs will not be routinely recorded]
   * Headache
   * Nausea (self-reporting; constructed questionnaire)
3. Patient treatment compliance (self-reporting; constructed questionnaire)
4. Clinical Pregnancy (positive BHCG and ultrasound evidence of fetal heart rate)

Study Design

Recruitment / Baseline Assessment The study population will be derived from a pool of patients referred to TCART (Toronto Centre for Assisted Reproductive Technology; Toronto, Canada). Patients that have been comprehensively evaluated for infertility and subsequently recommended to undergo controlled ovarian stimulation and intra-uterine insemination will be approached and recruited to participate in the study. Patients will be screened and evaluated for eligibility (based on the inclusion and exclusion criteria) by direct contact from one of the dedicated study investigators or dedicated research staff.

Randomization Randomization will be computer generated in a block design of 6 patients. Six corresponding opaque envelopes that enclose the blinded medication will be administered sequentially to consenting patients. Randomization will be performed at the start of the COH cycle and consequently the data will be analyzed as an intention-to-treat analysis.

Blinding Procedures Both patients and medical staff will be blinded to the treatment arms. Both the nimodipine (30 mg po qid) and placebo groups (placebo po qid) will receive 8 identical tablets with the same instructions for self-administration. The capsules will be only be identified by a unique study number to allow accurate analysis at the end of the study. A single pharmacy will be responsible for blinding, labeling and packaging the medication. Only the study coordinator (DN), who will not be involved clinically with study participants, will remain unblinded.

Interventions

Drug Formulation Nimotop® (Nimodipine) Bayer Pharmaceuticals Corporation. Calcium channel blocker. 30mg oral soft gelatin capsules.

Dosage Regimen Nimodipine is rapidly absorbed after oral administration reaching a peak concentration within one hour. It has a half-life of approximately 1-2 hours and a terminal clearance half-life of 8 hours, and thus requires relatively frequent administration. It is currently approved for the acute treatment of subarachnoid hemorrhage, with a dosing regimen of 60mg po q4h for 21 consecutive days. Several pharmacokinetic studies have focused on 30mg doses three times daily with no evidence of accumulation.

In our study intervention will be initiated once ovarian follicle maturation has been documented (≥1 ovarian follicle size of ≥ 17mm) and the absence of a premature LH surge has been confirmed - this will be classified as intervention day 0. Patients will receive oral nimodipine 30mg four times daily over a two day period with the following dosing schedule:

* Intervention Day 0 - noon / afternoon / bedtime (3 doses)
* Intervention Day 1 - morning / noon / afternoon / bedtime (4 doses)
* Intervention Day 2 - morning (1 dose)

Washout Period Nimodipine is eliminated almost exclusively in the form of metabolites. Less than 1% is recovered in the urine as unchanged drug. Over 95% of the medication is bound to plasma proteins. Nimodipine has a half life of 1-2 hours, with terminal elimination half life of approximately 8 hours. It should be completely eliminated from the body in about 40 hours.

Contraindications to Nimodipine use

* Hypersensitivity to the active substance or to any of the excipients of Nimodipine.
* The use of Nimodipine in combination with Rifampicin

Precautions to Nimodipine use

* Caution is required in patients with hypotension
* Nimodipine is metabolized by the cytochrome P450 3A4 system, therefore drugs (or grapefruit juice) that are known to either inhibit or to induce this enzyme should be taken into account, including:
* Rifampicin
* Quinupristin / Dalfopristin
* Valproic Acid
* Nortryptyline

Secondary Outcome variables:

* Side effects - Nausea, headache, lightheadedness, dizziness, diaphoresis, presyncopal or palpitations/tachycardia.
* Treatment compliance - Number of tablets taken (out of the prescribed 8 tablets), appropriate timing of medication (as instructed)
* Clinical pregnancy → positive bHCG serum test 2 weeks post IUI and ultrasound documentation of a fetal heart rate

Study - Delayed Ovulation Induction and Monitoring:

* Deviating from routine practice, our study protocol will call for a two-day delay in the hCG injection after the ultrasound detection of a mature ovarian follicle (intervention day 0). At this time point patients will have already been randomized and blinded to receive nimodipine 30 mg po qid, or placebo po qid for two days to ideally prevent the natural LH surge for a further 48 hours.
* During the two day period all study patients (nimodipine or placebo) will continue to be monitored daily at the clinic (mornings of day 1 and day 2) which will include transvaginal ultrasound and serum measurements of estradiol, LH and progesterone.
* If during the two day period an LH surge is detected during daily morning monitoring (eg. on day 1 or on day 2), the standard protocol of ovulation induction and IUI will be initiated - injection of hCG 250 mcg that same afternoon and two IUIs performed 16 hours and 40 hours after hCG injection. Participant will discontinue taking their assigned medication after an LH surge has been detected.
* If an LH surge is not detected during daily monitoring on day 1, the patient will continue taking their assigned medication and with daily monitoring.
* If an LH surge is not detected during daily monitoring by day 2, ovulation will be induced that same afternoon (~5 pm) by the injection of hCG 250 mcg followed by a single IUI 40 hours later.

Safety and Adverse Events Patients undergoing COS and IUI are regularly monitored for optimal treatment response and timing of IUI. Therefore investigators in this study will also have the opportunity to closely observe any safety or adverse events associated with the two-day duration of active intervention (nimodipine 30mg po qid x 48 hours). Specifically all patients will be asked about medication (nimodipine and placebo) compliance and side effects experienced during the morning cycle monitoring (day 1 and day 2).

Nimodipine has traditionally been investigated at higher does, frequencies and longer duration. According to the product monograph1, a dosing regimen of nimodipine 60mg po q4h resulted in the following side effects: hypotension (3.8%), nausea (1.2%), headache (1.2%) and bradycardia (1%). Conservative management consisted of discontinuing nimodipine and generally was effective in reversing the symptoms.

Data Analysis Plan / Statistical Plan Data will be expressed as mean +/- SD or percentage where applicable. Independent samples will be compared using the Student t test. The chi-squared test and Fisher exact test will be used for categorical data. A P value of <0.05 will be considered to indicate statistical significance.

Sample Size and Power Sample size calculations were performed using the computer program PS: Power and sample size calculation by William Dupont. We are planning a study of independent samples of treatments and controls with a 1:1 randomization. Expert opinion / prior data suggest that approximately 50% of patients in the placebo arm will have a natural LH surge detected on day 2 post intervention after a follicular maturation has been reached15. If 20% of patients in the nimodipine arm have a natural LH surge detected on day 2 post intervention, then we will need 38 subjects in each of the study arms to reject the null hypothesis (both groups have equal incidence of natural LH surge on day 2 post intervention) with a power of 0.8 and a type I error probability of 0.05. We anticipate approximately a 15% dropout rate leading to a total recruitment of 90 patients (45 per study arm).

ELIGIBILITY:
Inclusion Criteria: Infertility requiring intrauterine insemination

* Age: 25-40 (at time of enrollment)
* Intact Normal Ovaries (Both)
* Early follicular phase (day 2-4) serum FSH level < 20 mIU/ml
* Diagnosis of infertility with a recommended treatment of ovarian stimulation and IUI

Exclusion Criteria:

* BMI > 38 kg/m2
* Early follicular phase (day 2-4) serum FSH level ≥ 20 mIU/ml
* Overstimulated cycle: >3 mature follicles (≥17 mm)
* Abnormal uterine cavity and /or tubal blockage
* Diagnosis of infertility with a clear indication for IVF
* Severe male factor infertility: Total Motile Sperm Count < 2x106 post washing

Ages: 25 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2012-12; Primary Completion 2014-04 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Delay of LH surge by at least 2 days | From cycle day 3 until a spontaneous LH surge detected in the blood or the administration of the hCG trigger shot. Estimated time frame is 14 days.
  Nimodipine or placebo will be administered four times daily once the criterion for hCG triggering (one or more follicles at 1.7 cm diameter on ultrasound) is present in women being monitored for IUI.

SECONDARY OUTCOMES:
Side effect profile of nimodipine or placebo. | During tablet administration at mid-cycle.
  Any side effects (especially related to low blood pressure) will be reported by the subjects and recorded by the study investigators during the administration of nimodipine or placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Robert F Casper, MD, Principal Investigator — Toronto Centre for Advanced Reproductive Technology and University of Toronto
Locations (1):
- Toronto Centre for Advanced reproductive Technology (TCART), Toronto, Ontario, Canada

REFERENCES:
- [Background] Fainaru O, Firestone R, Casper RF. Oral nimodipine inhibits the ovarian cycle in mice. Fertil Steril. 2011 Mar 15;95(4):1494-6. doi: 10.1016/j.fertnstert.2010.12.008. Epub 2010 Dec 31. PMID 21195398